CLINICAL TRIAL: NCT01813968
Title: Ischemic Postconditioning in Cardiac Surgery
Acronym: IPICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Medical University of Warsaw (Other); University Hospital of North Norway (Other); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Mari-Liis Kaljusto, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/2613
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Surgery
Keywords: Ischemic postconditioning; Adult cardiac surgery; Aortic valve surgery; Swan-Ganz; Cardiac index
MeSH Terms: interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ischemic postconditioning (Experimental): Ischemic postconditioning via the cardioplegia line starting with 2 min of reperfusion followed by 2 min of "ischemia" x 3
  Interventions: Procedure: Ischemic postconditioning
- Control (No Intervention): Standard operating technique

INTERVENTIONS:
Procedure: Ischemic postconditioning
  Arms: Ischemic postconditioning

SUMMARY:
Ischemic postconditioning by repetitive cycles of reperfusion and ischemia has been proven both in animal models and in humans. This study aims to investigate the effect of ischemic postconditioning on postoperative hemodynamic function in a standard heart surgery patient population.

DETAILED DESCRIPTION:
Ischemic postconditioning is studied using cardiopulmonary bypass (CPB) and moderate hypothermia (32-34°C) in a patient population undergoing surgery of the aortic valve (repair/replacement ) or the ascending aorta. Postconditioning is applied by introducing reperfusion/ischemia via the cardioplegia line while the aorta is still cross-clamped thereby preventing the risk of additional neurological complications. All patients > 20 years eligible for aortic or aortic valve surgery and not affected by exclusion criteria, will be included.

The study is carried out as a randomised controlled multicenter study including 5-6 heart surgery centers.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective surgery of the ascending aorta or the aortic valve

-

Exclusion Criteria:

* Coronary artery disease requiring bypass surgery
* Tricuspid valve surgery
* Mitral valve surgery
* Atrial fibrillation (permanent or paroxysmal with or without concomitant ablation procedure)
* Patients on per oral or parenteral steroid therapy (inhalational steroids are allowed)
* Patients with autoimmune diseases
* "Redo" operations
* Active endocarditis (ongoing antibiotic therapy)
* On the discretion of the operating surgeon or anaesthesiologist

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2013-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Change in cardiac index between the groups during the first postoperative day | The first postoperative day: measurements at 2, 8 and 18 hrs postoperatively
  Cardiac index is measured by a Swan-Ganz catheter inserted preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery, Oslo University Hospital, Ullevål, Oslo, Norway